CLINICAL TRIAL: NCT07176065
Title: A Pilot Randomized Controlled Trial Assessing the Impact of Dexmedetomidine as an Adjunct to Periarticular Ropivacaine Infiltration on Postoperative Pain and Recovery in Patients Undergoing Total Knee Replacement
Brief Title: Dexmedetomidine as an Adjunct to Periarticular Ropivacaine in Total Knee Replacement: A Pilot Randomised Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ahmad Fariz Bin Elias, Clinical specialist, University of Malaya
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025429-15014
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain Management in Total Knee Arthroplasty
Keywords: Total Knee Replacement; TKR; Periarticular Infiltration; Ropivacaine; Dexmedetomidine; Postoperative Pain; Opioid Consumption; Regional Anaesthesia; Adductor Canal Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, quadruple-blinded randomised controlled trial. Sixty adult patients undergoing unilateral total knee replacement will be randomly assigned in a 1:1 ratio to receive periarticular infiltration with either ropivacaine alone (control group) or ropivacaine combined with 100 µg dexmedetomidine (intervention group). Allocation will be concealed using computer-generated block randomisation and sealed opaque envelopes. Blinding will be maintained for participants, care providers, investigators, and outcomes assessors. The intervention will be administered intraoperatively as a single dose.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be conducted in a quadruple-blinded manner. Group allocation will be concealed using computer-generated randomisation and sequentially numbered, opaque, sealed envelopes. A designated research team member, not involved in patient care or outcome assessment, will prepare the study drug (ropivacaine + saline or ropivacaine + dexmedetomidine) in identical, pre-labelled syringes. The operating surgeon, participant, and outcomes assessor will remain blinded to group allocation throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine + Saline (Active Comparator): Patients will receive 20 mL of periarticular infiltration consisting of 19 mL of 0.5% ropivacaine and 1 mL of normal saline during total knee replacement.
  Interventions: Drug: Ropivacaine + saline solution
- Ropivacaine + Dexmedetomidine (Experimental): Patients will receive 20 mL of periarticular infiltration consisting of 19 mL of 0.5% ropivacaine and 100 µg dexmedetomidine in 1 mL during total knee replacement.
  Interventions: Drug: Ropivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine + saline solution — 0.5% ropivacaine (19 mL) + 1 mL normal saline administered intraoperatively via periarticular injection.
  Arms: Ropivacaine + Saline
Drug: Ropivacaine + Dexmedetomidine — 0.5% ropivacaine (19 mL) + dexmedetomidine 100 µg in 1 mL administered intraoperatively via periarticular injection.
  Arms: Ropivacaine + Dexmedetomidine

SUMMARY:
This study aims to evaluate whether adding dexmedetomidine to ropivacaine-based periarticular infiltration (PAI) improves postoperative pain control in patients undergoing total knee replacement (TKR). Despite standard pain management, many patients continue to experience moderate-to-severe pain after surgery. Dexmedetomidine, a sedative and analgesic agent, may help prolong the effect of local anaesthetics. A total of 60 patients will be randomly assigned to receive either ropivacaine alone or ropivacaine with dexmedetomidine. Pain scores, opioid use, side effects, and recovery time will be monitored for 24 hours. The goal is to determine if this method is more effective and safer for improving recovery after knee surgery.

DETAILED DESCRIPTION:
Total knee replacement is associated with significant postoperative pain despite the use of multimodal analgesia. Periarticular infiltration (PAI) using local anaesthetics such as ropivacaine has become a common component of pain control protocols but offers a limited duration of relief. Dexmedetomidine, a selective α2-adrenergic agonist, has demonstrated analgesic benefits as an adjuvant in peripheral nerve blocks, but its role in PAI remains underexplored.

This double-blind randomised controlled trial will recruit 60 adult patients undergoing unilateral total knee replacement at Universiti Malaya Medical Centre. Patients will be randomly assigned to receive either PAI with 0.5% ropivacaine alone (control group) or ropivacaine combined with 100 µg dexmedetomidine (intervention group). All patients will receive spinal anaesthesia and an adductor canal block before surgery.

Pain scores will be recorded using the Numerical Rating Scale (NRS) at 1, 6, 12, and 24 hours postoperatively. Secondary outcomes include 24-hour opioid consumption (morphine milligram equivalents), patient satisfaction (5-point Likert scale), adverse effects (sedation, bradycardia, hypotension, PONV), and time to first ambulation. This study will provide important feasibility data and inform the design of a future multicentre trial, particularly within the Malaysian population.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Undergoing elective unilateral total knee replacement
* ASA physical status I-III
* No known allergy to local anaesthetics or dexmedetomidine
* No opioid use >24 hours preoperatively
* Provided informed consent

Exclusion Criteria:

* Known allergy to study drugs
* Chronic pain or neurological conditions
* Bilateral or revision TKR
* Significant deformity affecting function
* Substance abuse history
* Day-case surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
24-hour postoperative pain score (NRS 0-10) at rest and during movement | 24 hours postoperatively (from time of skin closure)
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates worst possible pain. Measurements will be taken at rest and during passive knee flexion to 90°, at 1, 6, 12, and 24 hours postoperatively. The primary endpoint is the NRS score at 24 hours.

SECONDARY OUTCOMES:
Total postoperative opioid consumption (MME) | 24 hours postoperatively
  Total opioid use in the first 24 hours postoperatively will be recorded from the PCA pump. All opioids will be converted into morphine milligram equivalents (MME) for standardisation.
Patient satisfaction with pain management | Postoperative day 1
  Patient satisfaction will be measured on postoperative day 1 using a 5-point Likert scale, ranging from "very dissatisfied" to "very satisfied."
Incidence of adverse effects (sedation, bradycardia, hypotension, PONV) | Within 24 hours postoperatively
  Adverse effects will be monitored and recorded within 24 hours postoperatively:
  Sedation (RASS ≤ -2) Bradycardia (HR < 50 bpm) Hypotension (MAP < 65 mmHg or SBP < 90 mmHg) PONV (score ≥1 on 0-4 scale)
Time to first ambulation | From end of surgery to first ambulation (within 24 hours)
  Time from skin closure to the patient's first unsupported ambulation (>5 metres) will be recorded in hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Protocol and statistical analysis plan
  Data collected from the study limited to demographic data, numerical rating scale and adverse event
Supporting Information: Study Protocol, SAP
Time Frame: 2 years after completing of study
Access Criteria: Editorial board that reviews my article for publication
  They will have assess to our data collection, as we will keep the data in redcap server
URL: https://redcap.um.edu.my/

REFERENCES:
- See also: We also register our research protocol to national medical research registration Malaysia — https://nmrr.gov.my/